CLINICAL TRIAL: NCT00613665
Title: Phase I, Randomized, Controlled, Single-blind, Dose-Ranging and Schedule-Finding Study of the Safety, Tolerability, and Immunogenicity of Chiron Helicobacter Pylori Vaccine in Healthy, Helicobacter Pylori-negative Adults
Brief Title: Safety and Immunogenicity of Chiron's Investigational H. Pylori Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HPP002
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Helicobacter Pylori; Gastritis; Gastric Cancer; Gastroduodenal Ulcers; Lymphoma
MeSH Terms: conditions — Gastritis; Stomach Neoplasms; Peptic Ulcer; Lymphoma

STUDY DESIGN:
Who Masked: Participant

ARMS (7):
- 1 (Experimental)
  Interventions: Biological: helicobacter pylori vaccine
- 2 (Experimental)
  Interventions: Biological: helicobacter pylori vaccine
- 3 (Experimental)
  Interventions: Biological: helicobacter pylori vaccine
- 4 (Experimental)
  Interventions: Biological: helicobacter pylori vaccine
- 5 (Placebo Comparator)
  Interventions: Biological: Placebo
- 6 (Experimental)
  Interventions: Biological: helicobacter pylori vaccine
- 7 (Experimental)
  Interventions: Biological: helicobacter pylori vaccine

INTERVENTIONS:
Biological: helicobacter pylori vaccine — Experimental H. pylori vaccine including NAP, CagA and VacA antigens (abbreviated HP3), 10 micrograms of each antigen, 0,1,2 month schedule (alum control was administered at 4 months), administered intramuscularly
  Arms: 1
Biological: helicobacter pylori vaccine — Seven subjects, experimental H. pylori vaccine including NAP, CagA and VacA antigens (abbreviated HP3), 25 micrograms of each antigen, 0,1,2 month schedule (alum control was administered at 4 months), administered intramuscularly
  Arms: 2
Biological: helicobacter pylori vaccine — Seven subjects, experimental H. pylori vaccine including NAP, CagA and VacA antigens (abbreviated HP3), 10 micrograms of each antigen, 0,1,4 month schedule (alum control was administered at 2 months), administered intramuscularly
  Arms: 3
Biological: helicobacter pylori vaccine — Eight subjects, experimental H. pylori vaccine including NAP, CagA and VacA antigens (abbreviated HP3), 25 micrograms of each antigen, 0,1,4 month schedule (alum control was administered at 2 months), administered intramuscularly
  Arms: 4
Biological: Placebo — Nine subjects, alum control (placebo comparator), 0,1,2,4 month schedule (served as control for arms 1-4), administered intramuscularly
  Arms: 5
Biological: helicobacter pylori vaccine — Nine subjects, experimental H. pylori vaccine including NAP, CagA and VacA antigens (abbreviated HP3), 10 micrograms of each antigen, 0,1,2 week schedule, administered intramuscularly
  Arms: 6
Biological: helicobacter pylori vaccine — Ten subjects, experimental H. pylori vaccine including NAP, CagA and VacA antigens (abbreviated HP3), 25 micrograms of each antigen, 0,1,2 week schedule, administered intramuscularly
  Arms: 7

SUMMARY:
This study was designed to investigate the safety and immunogenicity of Chiron's investigational H. pylori (HP3) vaccine

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Ages 18-40
* Negative for H. pylori infection
* Contraception for females

Exclusion Criteria:

* Present or past H. pylori infection
* Medically significant gastroduodenal disease
* Recent corticosteroid use
* Bleed diathesis
* Use of antibiotics used to treat H. pylori infection

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2001-02; Primary Completion 2001-12 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Safety measures: injection site and systemic reactions | 5 months

SECONDARY OUTCOMES:
Immunogencity measures: antigen-specific antibodies and cellular immune response | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Universitaetsklinikum Charité, Berlin, Germany